CLINICAL TRIAL: NCT00529048
Title: Quantification of the Incretin Effect in Healthy Subjects and Patients With Type 2 Diabetes Using Increasing Amounts of Oral Glucose Challenges
Brief Title: Quantification of the Incretin Effect in Healthy Subjects and Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: University of Copenhagen (Other); Merck Sharp & Dohme LLC (Industry); Forskningsrådet (Unknown); Diabetesforeningen (Other)
Responsible Party: Jonatan Bagger, University of Copehagen
Other Study IDs: INK-GLUKOSE1
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Incretin Effect
Keywords: Type 2 diabetes mellitus; Incretin effect; Glucagon-Like Peptide 1; Gastric Inhibitory Polypeptide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — p-Glucose p-Glucagon p-insulin p-c-pep. p-GLP-1 p-GIP Buffy coat s-paracetamol
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- T2DM: T2DM patients (WHO-criteria)
  Interventions: Other: Oral Glucose Tolerance Test; Other: Isoglycemic clamp; Other: Gastric emptying rate
- CTRL: Healthy control subjects matched individually to the cases.
  Interventions: Other: Oral Glucose Tolerance Test; Other: Isoglycemic clamp; Other: Gastric emptying rate

INTERVENTIONS:
Other: Oral Glucose Tolerance Test — The test is preformed 3 times with 3 different amounts of glucose (25g, 75g and 125g) deluded in 300ml of water.
Other: Isoglycemic clamp — I.v. glucose infusion initiating the glucose responds curves from the OGTT
Other: Gastric emptying rate — Paracetamol absorption test. Intake of 1,5g of paracetamol followed by measuring the absorption curve

SUMMARY:
Patients with T2DM lac a sufficient incretin response after oral glucose intake. It has only been tested using 50g of glucose. We don't know if patients with T2DM are capable of regulating the incretin effect like healthy people in responds to different amounts of glucose intake.

The aim of the present study is to quantify the incretin effect in healthy subjects and in patients with T2DM during increasing amounts of oral glucose challenges. The proposed studies will answer important questions on the mechanisms underlying T2DM and be of importance in relation to future preventive- and treatment strategies.

DETAILED DESCRIPTION:
The impaired incretin effect in patients with type 2 diabetes mellitus (T2DM) has previously only been evaluated using a glucose load of 50 g, and it is uncertain whether patients with T2DM are capable of regulating their incretin effect equivalent to healthy subjects. Furthermore, it is of great interest to quantify the secretion of GIP and GLP-1 during increasing glucose loads in both patients with T2DM and in healthy subjects in order to evaluate whether an increased secretion of one or both of the two incretin hormones contributes to the regulation of the incretin effect.

The aim of the present study is to quantify the incretin effect in healthy subjects and in patients with T2DM during increasing amounts of oral glucose challenges and corresponding isoglycemic iv glucose challenges. The proposed studies will answer important questions on the pathophysiology underlying T2DM and be of importance in relation to future preventive- and treatment strategies.

Eight patients with T2DM and 8 matched healthy subjects will be evaluated with oral glucose tolerance tests (OGTT) using increasing glucose loads (25, 50 and 100 g glucose) and isoglycemic iv glucose tolerance tests imitating the glucose concentrations as obtained during the oral glucose loads. The results will describe the regulation of the incretin effect in patients with T2DM and, thereby, contribute to the clarification of the pathophysiology of the postprandial hyperglycemia characterizing these patients.

ELIGIBILITY:
Inclusion Criteria: Cases

* Caucasians with T2DM according to WHO's criteria
* Normal Hemoglobin
* Agree to participate (orally and in writing)
* HbA1c: 6.5-9 %
* BMI: 23-35 kg/m2

Exclusion Criteria:Cases

* Liver disease (ALAT > 2 x normal level)
* Diabetic nephropathy (s-creatinin > 130 µM or albuminuria)
* Diabetic neuropathy (anamnestic)
* Proliferative diabetic retinopathy (anamnestic)
* Medical treatment witch cannot be stopped for 12 hours
* Pregnancy or breastfeed
* Treatment with Insulin or glitazones

Inclusion Criteria: Control group

* Caucasians
* Normal oral glucose tolerance according to WHO's criteria
* Normal Hemoglobin
* Agree to participate (orally and in writing)
* BMI: 23-35 kg/m2

Exclusion Criteria: Control group

* Liver disease (ALAT > 2 x normal level)
* Impaired function of the kidney (s-creatinin > 130 µM or albuminuria)
* Directly related til to someone suffering from diabetes mellitus
* Medical treatment witch cannot be stopped for 12 hours
* Pregnancy or breastfeed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Patients (Cases) will be recruted from the diabetes clinic at Depatment of Endocrinology at Herlev Hospital
  The control subjects will be recruted through the lokal papers, and individualy matched by age, sex and BMI to a patient befor enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2007-10; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Progress in Incretin effect in patients with T2DM compared with healthy subjects | 4 hours

SECONDARY OUTCOMES:
GIP and GLP-1 responscurvs | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tina Villsbøll, MD.DMSc., Study Chair — Herlev Hospital; Filip K Knop, MD.Phd., Study Director — Herlev Hospital
Locations (1):
- Endokrinologisk afd. J, Herlev Hospital, Herlev, Capital Region, Denmark

REFERENCES:
- [Background] Kolligs F, Fehmann HC, Goke R, Goke B. Reduction of the incretin effect in rats by the glucagon-like peptide 1 receptor antagonist exendin (9-39) amide. Diabetes. 1995 Jan;44(1):16-9. doi: 10.2337/diab.44.1.16. PMID 7813808
- [Background] Tseng CC, Zhang XY, Wolfe MM. Effect of GIP and GLP-1 antagonists on insulin release in the rat. Am J Physiol. 1999 Jun;276(6):E1049-54. doi: 10.1152/ajpendo.1999.276.6.E1049. PMID 10362617
- [Background] Wang Z, Wang RM, Owji AA, Smith DM, Ghatei MA, Bloom SR. Glucagon-like peptide-1 is a physiological incretin in rat. J Clin Invest. 1995 Jan;95(1):417-21. doi: 10.1172/JCI117671. PMID 7814643
- [Background] Habener JF. The incretin notion and its relevance to diabetes. Endocrinol Metab Clin North Am. 1993 Dec;22(4):775-94. PMID 8125072
- [Background] Edwards CM, Todd JF, Mahmoudi M, Wang Z, Wang RM, Ghatei MA, Bloom SR. Glucagon-like peptide 1 has a physiological role in the control of postprandial glucose in humans: studies with the antagonist exendin 9-39. Diabetes. 1999 Jan;48(1):86-93. doi: 10.2337/diabetes.48.1.86. PMID 9892226
- [Background] Gault VA, O'Harte FP, Harriott P, Mooney MH, Green BD, Flatt PR. Effects of the novel (Pro3)GIP antagonist and exendin(9-39)amide on GIP- and GLP-1-induced cyclic AMP generation, insulin secretion and postprandial insulin release in obese diabetic (ob/ob) mice: evidence that GIP is the major physiological incretin. Diabetologia. 2003 Feb;46(2):222-30. doi: 10.1007/s00125-002-1028-x. Epub 2003 Feb 12. PMID 12627321
- [Background] Miyawaki K, Yamada Y, Yano H, Niwa H, Ban N, Ihara Y, Kubota A, Fujimoto S, Kajikawa M, Kuroe A, Tsuda K, Hashimoto H, Yamashita T, Jomori T, Tashiro F, Miyazaki J, Seino Y. Glucose intolerance caused by a defect in the entero-insular axis: a study in gastric inhibitory polypeptide receptor knockout mice. Proc Natl Acad Sci U S A. 1999 Dec 21;96(26):14843-7. doi: 10.1073/pnas.96.26.14843. PMID 10611300
- [Background] Scrocchi LA, Brown TJ, MaClusky N, Brubaker PL, Auerbach AB, Joyner AL, Drucker DJ. Glucose intolerance but normal satiety in mice with a null mutation in the glucagon-like peptide 1 receptor gene. Nat Med. 1996 Nov;2(11):1254-8. doi: 10.1038/nm1196-1254. PMID 8898756
- [Background] Nauck M, Stockmann F, Ebert R, Creutzfeldt W. Reduced incretin effect in type 2 (non-insulin-dependent) diabetes. Diabetologia. 1986 Jan;29(1):46-52. doi: 10.1007/BF02427280. PMID 3514343
- [Background] Vilsboll T, Krarup T, Madsbad S, Holst JJ. Defective amplification of the late phase insulin response to glucose by GIP in obese Type II diabetic patients. Diabetologia. 2002 Aug;45(8):1111-9. doi: 10.1007/s00125-002-0878-6. Epub 2002 Jul 4. PMID 12189441
- [Background] Kjems LL, Holst JJ, Volund A, Madsbad S. The influence of GLP-1 on glucose-stimulated insulin secretion: effects on beta-cell sensitivity in type 2 and nondiabetic subjects. Diabetes. 2003 Feb;52(2):380-6. doi: 10.2337/diabetes.52.2.380. PMID 12540611
- [Background] Nauck MA, Homberger E, Siegel EG, Allen RC, Eaton RP, Ebert R, Creutzfeldt W. Incretin effects of increasing glucose loads in man calculated from venous insulin and C-peptide responses. J Clin Endocrinol Metab. 1986 Aug;63(2):492-8. doi: 10.1210/jcem-63-2-492. PMID 3522621
- [Background] Vilsboll T, Krarup T, Madsbad S, Holst JJ. Both GLP-1 and GIP are insulinotropic at basal and postprandial glucose levels and contribute nearly equally to the incretin effect of a meal in healthy subjects. Regul Pept. 2003 Jul 15;114(2-3):115-21. doi: 10.1016/s0167-0115(03)00111-3. PMID 12832099
- [Derived] Bagger JI, Knop FK, Lund A, Holst JJ, Vilsboll T. Glucagon responses to increasing oral loads of glucose and corresponding isoglycaemic intravenous glucose infusions in patients with type 2 diabetes and healthy individuals. Diabetologia. 2014 Aug;57(8):1720-5. doi: 10.1007/s00125-014-3264-2. Epub 2014 May 31. PMID 24879388
- [Derived] Bagger JI, Knop FK, Lund A, Vestergaard H, Holst JJ, Vilsboll T. Impaired regulation of the incretin effect in patients with type 2 diabetes. J Clin Endocrinol Metab. 2011 Mar;96(3):737-45. doi: 10.1210/jc.2010-2435. Epub 2011 Jan 20. PMID 21252240